CLINICAL TRIAL: NCT03680053
Title: A Randomized Comparison of the Live Birth Rate Between the Progestin-primed Ovarian Stimulation Protocol and the Gonadotrophin Releasing Hormone Antagonist Protocol in Patients Undergoing in Vitro Fertilization
Brief Title: Comparison of the Live Birth Rate Between the PPOS and the GnRH Antagonist Protocol in Patients Undergoing IVF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to difficulty in recruiting patients.
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIAI 2018-08
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-08

CONDITIONS: Infertility; ART
MeSH Terms: conditions — Infertility | interventions — Dydrogesterone; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPOS group (Experimental): Ovarian stimulation will use the progestin-primed ovarian stimulation (PPOS) protocol.Women will receive progesterone (oral duphaston 20mg) daily from Day 3 till the day of ovulation trigger.
  Interventions: Drug: Duphaston
- Antagonist group (Active Comparator): Ovarian stimulation will use the antagonist protocol. Women will receive antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.
  Interventions: Drug: Cetrorelix

INTERVENTIONS:
Drug: Duphaston — Women will receive oral duphaston 20mg daily from Day 3 till the day of ovulation trigger.
  Arms: PPOS group
Drug: Cetrorelix — Women will receive antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.
  Arms: Antagonist group

SUMMARY:
A randomized comparison of the live birth rate between the progestin-primed ovarian stimulation protocol and the gonadotrophin releasing hormone antagonist protocol in patients undergoing in vitro fertilization

Research question Does the live birth rate of the progestin-primed ovarian stimulation protocol comparable with the GnRH antagonist protocol for patients undergoing IVF?

Design This is a randomized controlled trial.

Research plan

Population: Infertile women who have medical indication for IVF will be recruited for study if they fulfil the selection criteria.

Intervention: Women will receive oral dydrogesterone 20mg daily from Day 3 till the day of ovulation trigger.

Comparator: Women will receive antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.

Outcomes: The primary outcome is the live birth rate the first FET.

Ovarian stimulation, egg retrieval, embryos frozen and frozen embryo transfer will be performed according to the standard operating procedures of the centres.

ELIGIBILITY:
Inclusion Criteria:

* Age of women <43 years at the time of ovarian stimulation for IVF
* Antral follicle count (AFC) on day 2-5 of the period≥5

Exclusion Criteria:

* Presence of a functional ovarian cyst with E2>100 pg/mL
* Recipient of oocyte donation
* Undergoing preimplantation genetic testing
* Presence of hydrosalpinx which is not surgically treated or endometrial polyp on scanning during ovarian stimulation

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
live birth rate of the first FET live birth rate of the first FET live birth rate | a live birth after 22 weeks gestation, through study completion, an average of 1 year
  live birth rate of the first FET

SECONDARY OUTCOMES:
Serum estradiol level | on the day of hCG trigger, an average of 2 weeks after randomization
  Serum estradiol level on the day of hCG trigger
Serum progesterone level | on the day of hCG trigger, an average of 2 weeks after randomization
  Serum progesterone level on the day of hCG trigger
Serum LH level | on the day of hCG trigger, an average of 2 weeks after randomization
  Serum LH level on the day of hCG trigger
Serum FSH level | on the day of hCG trigger, an average of 2 days after randomization
  Serum FSH level on Day 2 of the period
oocyte retrieved number | the number of oocyte retrieved, an average of 2 weeks after randomization
embryo number | the number of embryo, an average of 3 weeks after randomization
positive hCG level | a blood hCG test is performed 14 days after the FET, up to 14 days
  defined with the result of serum β-hCG ≥10 mIU/mL
clinical pregnancy rate | presence of intrauterine gestational sac on ultrasound at 6 weeks of pregnancy, up to 6 weeks
  presence of intrauterine gestational sac on ultrasound at 6 weeks of pregnancy
ongoing pregnancy rate | viable pregnancy beyond gestation 12 weeks, up to 12 weeks
  presence of a fetal pole with pulsation at 12 weeks of gestation
implantation rate | number of gestational sacs per embryo transferred at 6 weeks of pregnancy, up to 6 weeks
  number of gestational sacs per embryo transferred
multiple pregnancy rate | multiple pregnancy beyond gestation 12 weeks up to 12 weeks
  more than one intrauterine sacs on scanning
miscarriage rate | a clinically recognized pregnancy loss before the 22 weeks of pregnancy, up to 22 weeks
  defined as a clinically recognized pregnancy loss before the 22 weeks of pregnancy. The denominator is the clinical pregnancy.
ectopic pregnancy rate | ectopic pregnancy during first trimester, up to 12 weeks
  pregnancy outside the uterine cavity
birth weight | a live birth after 22 weeks gestation, through study completion, an average of 1 year
  birth weight of the baby delivered
rate of participants with adverse events | adverse events during COH in an average of 1 month
  adverse events during COH
rate of obstetric complications | obstetric complications during pregnancy or delivery in an average of 1 year
  obstetric complications during pregnancy or delivery. The information will be acquired by contacting all the participants through phone
rate of fetal or congenital defects | fetal or congenital defects found during pregnancy or delivery in an average of 1 year
  fetal or congenital defects found during pregnancy or delivery. The information will be acquired by contacting all the participants through phone

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Principal Investigator — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- ShangHai JIAI Genetics&IVF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared. Data will be available when beginning 3 months and ending 5 years following article publication. To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with.Data will be made available by the following way. Proposals should be directed to lihe198900@163.com. And data are available for 5 years at a third party website (link to be included after the article publication).
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Al-Inany HG, Youssef MA, Aboulghar M, Broekmans F, Sterrenburg M, Smit J, Abou-Setta AM. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2011 May 11;(5):CD001750. doi: 10.1002/14651858.CD001750.pub3. PMID 21563131
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Dong J, Wang Y, Chai WR, Hong QQ, Wang NL, Sun LH, Long H, Wang L, Tian H, Lyu QF, Lu XF, Chen QJ, Kuang YP. The pregnancy outcome of progestin-primed ovarian stimulation using 4 versus 10 mg of medroxyprogesterone acetate per day in infertile women undergoing in vitro fertilisation: a randomised controlled trial. BJOG. 2017 Jun;124(7):1048-1055. doi: 10.1111/1471-0528.14622. PMID 28276192
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975